CLINICAL TRIAL: NCT01626313
Title: UCLA FOCUS (Families OverComing Under Stress) Family Resiliency Training Research Study
Brief Title: UCLA FOCUS Family Resiliency Training Research Study
Acronym: FOCUS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Proposed studies were not funded
Sponsor: University of California, Los Angeles (Other)
Collaborators: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Shirley Glynn, Associate Researcher, University of California, Los Angeles
Allocation: Randomized | Masking: None | Purpose: Supportive Care
Other Study IDs: 11-003001
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Veteran Families; Family Communications; Civilian Life Reintegration
Keywords: Veteran families; OEF; OIF; OND; Resiliency; Psycho educational training; Stress; Military

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate intervention (Active Comparator): Subjects are randomized to receive immediate intervention of the 8 session FOCUS IFRT
  Interventions: Behavioral: FOCUS Individualized Family Resiliency Training
- Waitlisted (Active Comparator): Subjects are randomized to be waitlisted for 4 months, re-assessed and then receive intervention of the 8 session FOCUS IFRT
  Interventions: Behavioral: FOCUS Individualized Family Resiliency Training

INTERVENTIONS:
Behavioral: FOCUS Individualized Family Resiliency Training — Eight session psycho educational training for families to enhance communication and reduce stressors related to return to post-military life.

SUMMARY:
The study will examine the effectiveness of an eight session, manualized individual family resiliency training (IFRT) for families with one OEF/OIF/OND veteran in promoting better family communication relating to return to post military life.

ELIGIBILITY:
Inclusion Criteria:

* OEF/OIF/OND Veteran adult family member
* cohabiting with significant other for 6 months or more
* at least one child age 5 to 17 years

Exclusion Criteria:

* active case with Child Protective Services
* conditions or substance use that limits ability to fully participate in the research program

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12 (Estimated); Primary Completion 2013-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Improvement on standardized behavioral health assessment scales | 4-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Patricia E Lester, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Semel Institute, Los Angeles, California, United States